CLINICAL TRIAL: NCT01731145
Title: Quantitative Assessment of Tremor Using Portable Six-axis (Tri-axial Accelerometer and Tri-axial Gyroscope) Motion Sensing System
Brief Title: Assessment of Tremor Using SNUMAP Motion Sensing System
Acronym: SNUMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Life Science Technology Inc. (Industry)
Responsible Party: Principal Investigator, BS Jeon, Professor and Chairman, Department of Neurology, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D-1407-011-590
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Tremor
Keywords: Tremor; SNUMAP; accelerometry; gyroscope; clinical rating scale
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SNUMAP assessment (Experimental): Uses SNUMAP motion sensing system to quantify tremor symptom.
  Interventions: Device: SNUMAP

INTERVENTIONS:
Device: SNUMAP — Portable six-axis (tri-axial accelerometer and tri-axial gyroscope) motion sensing system
  Other Names: Hybrid (accelerometer and gyroscope)

SUMMARY:
The purpose of this study is to record and measure tremor using portable six-axis (tri-axial accelerometer and tri-axial gyroscope) motion sensing system.

DETAILED DESCRIPTION:
SNUMAP system is portable, finger-worn, battery powered device that contains MEMS (micro-electro-mechanical system) hybrid motion sensor (three-axis accelerometer and three-axis gyroscope). The SNUMAP device consists of a wrist module and finger module, which attaches to an patients's finger and transmits three dimensional motions to a wrist module for storage and further analysis. The aims of this study is to assess tremor severity using tri-axial accelerometry and gyroscope to determine the reliability and the correlation with clinical measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-80 years
* Patients with tremor (involuntary, rhythmic, oscillatory movement in one or more body part)
* Subject who signed an informed consent

Exclusion Criteria:

* Pregnant or nursing woman.
* Comorbid neurologic illnesses that impact the ability to perform the study tasks.
* Subjects with medical condition that in the opinion of the investigator would affect his/her ability to participate in this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
3-D Accelerometric and gyroscope variables measured | 1 day
  Correlation between SNUMAP motion sensing system symptom assessment and clinical tremor rating scale (TRS) scores

CONTACTS AND LOCATIONS:
Overall Officials: Beom S Jeon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Neurology, Seoul National University Hospital, Seoul, South Korea